CLINICAL TRIAL: NCT01643005
Title: Pilot Phase of Couples-Based Intervention to Reduce HIV/STD Risk (Concurrency, Number of Partners, Unprotected Sex), Strengthen Relationships, and Improve Parenting Among Young Parenting Heterosexual Couples
Brief Title: A Couple-Based Relationship Strengthening HIV Intervention for Young Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1105008508; R34MH094354 (NIH)
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: HIV
Keywords: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Control Group (Active Comparator): For the active control group we will use Nurturing Parenting Groups currently being run by the community collaborator.
  Interventions: Behavioral: Parenting Program Intervention
- Relationship Strengthening HIV Prevent. (Experimental): The relationship strengthening HIV intervention will build on the structure of the Nurturing Parenting Groups and will be integrated so that participants will receive the Nurturing Parenting Groups plus the relationship strengthening HIV intervention.
  Interventions: Behavioral: Relationship Strengthening HIV Prevention Intervention

INTERVENTIONS:
Behavioral: Relationship Strengthening HIV Prevention Intervention — The relationship strengthening HIV intervention will build on the structure of the Nurturing Parenting Groups and will be integrated so that participants will receive the Nurturing Parenting Groups plus the relationship strengthening HIV intervention.
  Other Names: Partners in Life
  Arms: Relationship Strengthening HIV Prevent.
Behavioral: Parenting Program Intervention — Nurturing Parenting curriculum delivered in a group format.
  Other Names: Nurturing Parenting
  Arms: Active Control Group

SUMMARY:
This study seeks to develop, implement, and assess an innovative 15-session couple-based intervention to be delivered in a group format to young parents that aims to strengthen relationships and reduce HIV risk. The ultimate goal of our intervention is to reduce HIV/STD risk (concurrency, number of partners, unprotected sex), strengthen relationships, and improve parenting among young parenting heterosexual couples.

DETAILED DESCRIPTION:
This study develops a couple-based HIV prevention intervention that is innovative and important because it integrates an intervention that improves sexual health, relationship functioning, and parenting skills. Our intervention will be integrated with an existing community based parenting program. By targeting high risk heterosexual couples experiencing an important life transition that increases their stress, conflict, and sexual risk, the investigators can provide maximum benefit to the men, women, and children in our communities. Using the guiding framework of Attachment Theory and the principles of Emotion Focused Therapy, the investigators will directly address issues of emotion, intimacy,and relationship functioning to create an intervention that strengthens romantic relationships and reduces HIV risk behavior. The investigators will conduct a small pilot randomized controlled trial of 50 parenting couples randomized to either the relationship strengthening HIV prevention intervention or an active control. The intervention will last 15 weeks and each session will be approximately 1.5 hours long. The investigators will assess couples at baseline, 4-months, and 8-months.

ELIGIBILITY:
Inclusion Criteria:

* Women's age between 14 and 25
* Men's age 14 or older
* Have a child that is 0-1 year old
* In a romantic relationship with the mother/father of the baby
* Not known to be HIV positive
* English speaking

Exclusion Criteria:

* Child older than 1 year
* HIV positive

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-08; Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
High risk sexual behavior | Baseline
  Number of sexual partners, Concurrent sexual partners, Unprotected sex, Repeat pregnancy
High risk sexual behavior | 4 months
  Number of sexual partners, Concurrent sexual partners, Unprotected sex, Repeat pregnancy
High risk sexual behavior | 8 months
  Number of sexual partners, Concurrent sexual partners, Unprotected sex, Repeat pregnancy

SECONDARY OUTCOMES:
Relationship Functioning at 4 months | 4 months
Relationship Dissolution at 4 months | 4 months
Change from Baseline in relationship based determinants at 4 months | 4 months
  Attachment, Intimacy, Communication, Equity, Relationship Conflict
Relationship Functioning at 8 months | 8 months
Relationship Dissolution at 8 months | 8 months
Change from Baseline in relationship based determinants at 8 months | 8 months
  Attachment, Intimacy, Communication, Equity, Relationship Conflict

CONTACTS AND LOCATIONS:
Overall Officials: Trace S Kershaw, PhD, Principal Investigator — Yale School of Public Health
Locations (1):
- Children's Community Programs of Connecticut, New Haven, Connecticut, United States